CLINICAL TRIAL: NCT04164680
Title: Relationship Between Simultaneously Acquired Resting-state Regional Cerebral Glucose Metabolism and Functional MRI in DOC: a PET/MR Hybrid Scanner Study
Brief Title: Simultaneously PET/MRI in Prolonged DOC Patients
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Dr., Hangzhou Normal University
Other Study IDs: 2019N55749
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Disorder of Consciousness; Minimally Conscious State; FDG-PET; Rs-fMRI
Keywords: Disorder of Consciousness; Unresponsive wakefulness syndrome; Multimodal Neuroimaging
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with disorders of consciousness
  Interventions: Diagnostic Test: Multimodal Neuroimaging

INTERVENTIONS:
Diagnostic Test: Multimodal Neuroimaging — fludeoxyglucose (FDG-)PET/MR imaging

SUMMARY:
Recently introduced hybrid PET/MR scanners provide the opportunity to measure simultaneously, and in direct spatial correspondence, both metabolic demand and functional activity of the brain, hence capturing complementary information on the brain's physiological state. Here we exploited PET/MR simultaneous imaging to explore the relationship between the metabolic information provided by resting-state fluorodeoxyglucose-PET (FDG-PET) and fMRI (rs-fMRI) in patients with disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* DOC patients （acute, subacute or chronic period）: Coma, UWS and MCS.

Exclusion Criteria:

* neuromuscular blocking agents or sedative drugs administered within the prior 24 hours；
* unstable medical condition；
* mental implant in the brain

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Distinguishing patients in unresponsive wakefulness syndrome, UWS [i.e. patients showing eyes opening but no behavioral evidence of consciousness ] from patients in minimally conscious state, MCS [i.e., patients showing minimal, inconsistent but clearly discernible intentional behaviors ] is pivotal for decision making in the entire care pathway of patients with DoC.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
resting-state fMRI | Within 7 days
  Use resting-state fMRI to test the functional connectivity
fludeoxyglucose (FDG-)PET | Within 7 days
  UseFDG-PET to test the metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Cavaliere C, Kandeepan S, Aiello M, Ribeiro de Paula D, Marchitelli R, Fiorenza S, Orsini M, Trojano L, Masotta O, St Lawrence K, Loreto V, Chronik BA, Nicolai E, Soddu A, Estraneo A. Multimodal Neuroimaging Approach to Variability of Functional Connectivity in Disorders of Consciousness: A PET/MRI Pilot Study. Front Neurol. 2018 Oct 18;9:861. doi: 10.3389/fneur.2018.00861. eCollection 2018. PMID 30405513